CLINICAL TRIAL: NCT07160933
Title: Adaptation and Refinement of a Psychosocial Intervention to Reduce Post-Traumatic Stress in Young Adult Survivors of Cancer
Brief Title: Development of a Psychosocial Intervention to Reduce Post Traumatic Stress in Young Adult Survivors of Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zeba Ahmad, Ph.D. (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor-Investigator, Zeba Ahmad, Ph.D., Clinical Staff Psychologist, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-306; CSDG-24-1319592-01-CTPS (Other Grant/Funding Number: American Cancer Society Clinician Scientist Development Grant (CSDG))
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-09

CONDITIONS: Post-traumatic Stress Symptoms
Keywords: young adult cancer survivors; cancer-related post-traumatic stress; post-traumatic stress
MeSH Terms: interventions — Psychosocial Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psychosocial Intervention for Cancer-Related Post-Traumatic Stress in Young Adults (Experimental): The study team aims to evaluate the feasibility and acceptability of the adapted psychosocial intervention through a pilot trial with a group of 80 YACs, followed by mixed-methods data analysis of feasibility and acceptability outcomes.
  Interventions: Behavioral: Psychosocial Intervention for Cancer-Related Post-Traumatic Stress in Young Adults

INTERVENTIONS:
Behavioral: Psychosocial Intervention for Cancer-Related Post-Traumatic Stress in Young Adults — A new group-based virtual intervention to address post-traumatic stress related to cancer in YACs, integrating evidence-guided treatments from Cognitive Processing Therapy and Mind-Body Resiliency interventions.

SUMMARY:
The goal of this study is to develop a virtual group intervention to address post-traumatic stress related to cancer in young adult cancer survivors (YACs, aged 18-39). The study team will do this by integrating evidence-guided treatments and expert clinician feedback (N=10) on the content, delivery, and structure of the intervention. Next, the study team will refine this intervention through a pilot trial with a group of YACs (N=80).

ELIGIBILITY:
Inclusion Criteria: To be eligible for this study, participants will be:

* Currently aged between 18 - 39;
* Currently receiving or having completed treatment for cancer at the Mass General Cancer Institute within the past 5 years;
* Reporting a score denoting at least mild symptoms of PTSD on the Post-traumatic Stress Checklist 5 (PCL-5);
* English-speaking;
* Have access to a device with audio/video capabilities to complete virtual intervention sessions.

Exclusion Criteria:

* Unable to provide verbal consent
* Reporting active symptoms of psychosis that preclude safe participation.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-16 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Intervention Feasibility: Percent of Identified Prospective Participants Who Enroll | Post-treatment completion (enrollment to treatment completion is approximately 3 months)
  Percent of eligible participants who were offered participation and who enroll in the study by completing consent and baseline assessment.
Intervention Feasibility: Proportion of Participants Completing the Program | Post-treatment completion (enrollment to treatment completion is approximately 3 months)
  Percent of enrolled participants who complete the program, defined as completing 6 out of 8 sessions.
Intervention Acceptability | Post-treatment completion (enrollment to treatment completion is approximately 3 months)
  Acceptability will be assessed by the Client Satisfaction Questionnaire (CSQ-8). The intervention study will be considered acceptable if ≥80% of participants rate it as acceptable (defined as a CSQ-8 score ≥20).

CONTACTS AND LOCATIONS:
Locations (1):
- Mass General Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No